CLINICAL TRIAL: NCT04640077
Title: Donanemab Follow-On Study: Safety, Tolerability, And Efficacy in Symptomatic Alzheimer's Disease With Validation of Remote Neuropsychological Assessments
Brief Title: A Follow-On Study of Donanemab (LY3002813) With Video Assessments in Participants With Alzheimer's Disease (TRAILBLAZER-EXT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17447; I5T-MC-AACH (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Cognitive Dysfunction | interventions — donanemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Validation of Remote Scale Assessments (Other): Participants from the originating trials did not receive any drug in Part A. Participants were randomized 1:1 into two groups to have their cognitive and functional scales assessed.
  Group 1: Cognitive/functional scale assessment at the study site (on-site), followed by an at-home assessment (VTC; video teleconference), or Group 2: Cognitive/functional scale assessment at home (VTC), followed by assessment on-site.
  Total time in Part A was up to 24 weeks.
  Interventions: Other: No Intervention
- Part B: Donanemab (Experimental): Participants who had received placebo in the originating trials received 700 milligrams (mg) donanemab administered intravenously (IV) every 4 weeks (Q4W) for 3 doses, then 1400 mg donanemab administered IV Q4W for up to 48 weeks.
  Interventions: Drug: donanemab

INTERVENTIONS:
Other: No Intervention — No intervention
  Arms: Part A: Validation of Remote Scale Assessments
Drug: donanemab — Administered IV
  Other Names: LY3002813
  Arms: Part B: Donanemab

SUMMARY:
The main goals of this study are to further determine whether the study drug donanemab is safe and effective in participants with Alzheimer's disease and to validate neuropsychological assessments administered over videoconferencing

ELIGIBILITY:
Inclusion Criteria:

* Participated in a double-blind treatment period of a sponsor-approved originating donanemab trial, for example the TRAILBLAZER-ALZ study.
* Have a study partner
* Stable symptomatic Alzheimer's Disease (AD) medications and other medication that may impact cognition for at least 30 days prior to randomization into Part A

Exclusion Criteria:

* Current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with outcome assessments or the analyses in this study.
* Have received treatment with a passive anti-amyloid immunotherapy after completion of originating donanemab study or received active immunization against Aβ in any other study.
* Poor venous access
* Contraindication to PET or MRI imaging

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (23):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - UC Irvine-Institute for Memory Impairments and Neurological Disorders (UCI MIND), Irvine, California
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Synexus Clinical Research US, Inc., Orlando, Florida
  - Advanced Research Consultants, Palm Beach Gardens, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group - Hyde Park, Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - The University of Kansas - Clinical Research Center, Fairway, Kansas
  - Cotton O'Neil Clinical Research Center - Central Office, Topeka, Kansas
  - Boston Center for Memory, Newton, Massachusetts
  - Washington University, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Guilford Neurologic Research, PA, Greensboro, North Carolina
  - Ohio State University, Columbus, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Abington Neurological Associates, Ltd., Abington, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - National Clinical Research, Inc, Richmond, Virginia
- Canada (4):
  - Bruyère Research Institute, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Clinique de la Mémoire de l'Outaouais, Gatineau, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: Access Criteria:
  A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Follow-On Study of Donanemab (LY3002813) With Video Assessments in Participants With Alzheimer's Disease (TRAILBLAZER-EXT) — https://trials.lillytrialguide.com/en-US/trial/7tATxSc3LHXNDE2nVmdIY

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study AACH was an extension of sponsor-approved originating donanemab studies AACC (NCT01837641) and AACG (NCT03367403). This was a two-part study (Parts A and B). Participants received the study drug only in Part B, whereas Part A consisted of clinical assessments.
Pre-assignment Details: Participants in Part A were randomized 1:1 into two groups (Group 1 and Group 2) to have their cognitive and functional scales assessed.
Groups:
- Part A - Group 1: Validation of Remote Scale Assessments: Participants from the originating trials did not receive any drug in Part A.
  Participants in Group 1 underwent cognitive/functional scale assessment at the study site (on-site), followed by an at-home assessment (VTC; video teleconference).
  Total time in Part A - Group 1 was up to 24 weeks.
- Part A - Group 2: Validation of Remote Scale Assessments: Participants from the originating trials did not receive any drug in Part A.
  Participants in Group 2 underwent cognitive/functional scale assessment at home (VTC), followed by assessment on-site.
  Total time in Part A - Group 2 was up to 24 weeks.
Period: Period 1
Arm/Group | Part A - Group 1: Validation of Remote Scale Assessments | Part A - Group 2: Validation of Remote Scale Assessments | Part B: Donanemab
Started | 50 | 45 | 0
Received At Least 1 Dose of Study Drug | 0 | 0 | 0
Completed | 43 | 39 | 0
Not Completed | 7 | 6 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Screen Failure | 2 | 0 | 0
Period: Period 2
Arm/Group | Part A - Group 1: Validation of Remote Scale Assessments | Part A - Group 2: Validation of Remote Scale Assessments | Part B: Donanemab
Started | 0 | 0 | 55 (After Part A, participants who had received placebo in the originating trials moved to Part B.)
Received At Least 1 Dose of Study Drug | 0 | 0 | 55
Completed | 0 | 0 | 25
Not Completed | 0 | 0 | 30
Not completed — Withdrawal by Subject | 0 | 0 | 18
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Death | 0 | 0 | 2
Not completed — Progressive Disease | 0 | 0 | 1
Not completed — Withdrawal Due To Caregiver Circumstances | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants in Part A.
Groups:
- Part A: Validation of Remote Scale Assessments: Participants from the originating trials did not receive any drug in Part A. Participants were randomized 1:1 into two groups to have their cognitive and functional scales assessed.
  Group 1: Cognitive/functional scale assessment at the study site (on-site), followed by an at-home assessment (VTC; video teleconference), or Group 2: Cognitive/functional scale assessment at home (VTC), followed by assessment on-site.
  Total time in Part A was up to 24 weeks.
  After Part A, participants who had received placebo in the originating trials moved to Part B.
Arm/Group | Part A: Validation of Remote Scale Assessments
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 93
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Part A: Intraclass Correlation Between On-Site and Video Teleconference (VTC) Assessments
Description: Part A didn't involve any drug and drug related efficacy analyses. Participants in Part A were divided into 2 groups, and they completed the same set of clinical assessments. Participants in Part A Group 1 completed the clinical assessments at a clinic site first (on-site) followed by at home assessments (VTC). Participants in Part A Group 2 completed the assessments at home first, followed by on-site assessment. The goal of Part A was to evaluate the comparability of remote and on-site clinical assessments. The intra-class correlation coefficient (ICC), a measure of agreement for continuous outcome measures, was used to determine agreement between remote and onsite assessments for each outcome measure. Outcome measure tested were the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog13), Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (ADCS-ADL), Mini Mental State Examination (MMSE), and Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB).
Time Frame: Baseline to 4 Weeks
Population: All participants in Part A who had evaluable data for this outcome.
Measure: Number (95% Confidence Interval); unit: Intraclass correlation coefficient
Groups:
- Part A: Validation of Remote Scale Assessments: Participants from the originating trials did not receive any drug in Part A. Participants were randomized 1:1 into two groups to have their cognitive and functional scales assessed.
  * Group 1: Cognitive/functional scale assessment at the study site (on-site), followed by an at-home assessment (VTC; video teleconference), or
  * Group 2: Cognitive/functional scale assessment at home (VTC), followed by assessment on-site.
Arm/Group | Part A: Validation of Remote Scale Assessments
Number analyzed (Participants) | 84
Intraclass correlation coefficient
  ADAS-Cog13: number analyzed (Participants) | 81
  ADAS-Cog13 | 0.8172 [0.7293 to 0.8785]
  ADCS-ADL: number analyzed (Participants) | 82
  ADCS-ADL | 0.8819 [0.8227 to 0.9222]
  MMSE | 0.8251 [0.7148 to 0.8907]
  CDR-SB: number analyzed (Participants) | 80
  CDR-SB | 0.8254 [0.7380 to 0.8852]

2. Primary Outcome: Part B: Percentage of Participants With One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Percentage of participants with TEAEs and SAEs were reported here. A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this record.
Time Frame: Baseline Up To 96 Weeks
Population: All participants from Part B, who received at least one dose of donanemab.
Measure: Number; unit: Percentage of participants
Groups:
- Part B: Donanemab: Participants who had received placebo in the originating trials received 700 mg donanemab administered IV Q4W for 3 doses, then 1400 mg donanemab administered IV Q4W for up to 48 weeks.
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
Percentage of participants
  TEAEs | 90.9
  SAEs | 29.1

3. Primary Outcome: Part B: Number of Participants With Suicidality Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Number of Participants with Suicidality Based on C-SSRS was reported.
Time Frame: Baseline, Week 72
Population: All participants in Part B, who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 53
Participants
  Suicidal Ideation | 3
  Suicidal Behavior | 1

4. Secondary Outcome: Part B: Change From Baseline on the Mini Mental State Examination (MMSE) Score
Description: The MMSE is an instrument used to assess cognitive function in participants. The instrument measures orientation, memory, and attention; the ability of the participant to name objects; follow verbal and written commands; write a sentence; and copy figures. The range for the total MMSE score is 0 to 30, with lower scores indicating greater level of impairment. LS Mean was determined by Mixed Models for Repeated Measurements (MMRM) model with Baseline + Visit + Baseline*Visit + Age + Years of Education + Presence/ Absence of Anti-dementia Drugs as variables.
Time Frame: Baseline, Week 72
Population: All participants in Part B who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
Score on a scale | -0.87 (0.557)

5. Secondary Outcome: Part B: Change From Baseline on the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) Score
Description: The ADAS-Cog13 (13-item version of ADAS Cog) assesses areas of cognitive function that are the most typically impaired in Alzheimer's Disease (AD): orientation, verbal memory, language, praxis, delayed free recall, digit cancellation, and maze-completion measures. The ADAS-Cog13 scale ranges from 0 to 85, with higher scores indicating greater disease severity. LS Mean was determined by MMRM model with Baseline + Visit + Baseline*Visit + Age + Years of Education + Presence/Absence of Anti-dementia Drugs as variables.
Time Frame: Baseline, Week 72
Population: All participants in Part B, who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
Score on a scale | 4.63 (1.195)

6. Secondary Outcome: Part B: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS)
Description: The iADRS is a composite that measures both cognition and function from the ADAS-Cog and the ADCS-iADL (Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living). The iADRS is calculated as a linear combination of the total scores of the ADAS-Cog13 (score range 0 to 85 with higher scores reflecting worse performance) and the ADCS-iADL (score range from 0-59 with higher scores reflecting better performance). The iADRS score ranges from 0 to 144 with lower scores indicating greater impairment. LS Mean was determined by MMRM model using Baseline + Visit + Baseline*Visit + Age + Years of Education + Presence/Absence of Anti-dementia Drugs as variables.
Time Frame: Baseline, Week 72
Population: All participants in Part B, who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
Score on a scale | -10.14 (1.850)

7. Secondary Outcome: Part B: Change From Baseline on the Alzheimer's Disease Cooperative Study - Instrumental Activities of Daily Living (ADCS-iADL)
Description: The ADCS-iADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean was determined by MMRM model using = Baseline + Visit + Baseline*Visit + Age + Years of Education + Presence/Absence of Anti-dementia Drugs as variables.
Time Frame: Baseline, Week 72
Population: All participants in Part B, who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
Score on a scale | -6.21 (1.149)

8. Secondary Outcome: Part B: Change From Baseline on the Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB)
Description: The CDR-SB is a global assessment tool than can be used to effectively evaluate both cognition and function. Participant's cognitive status is rated across 6 domains or 'boxes' of functioning: Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care. The CDR-SB scores are calculated by adding the box scores and range from 0 to 18 with higher scores indicative of more impairment. LS Mean was determined by MMRM model using Baseline + Visit + Baseline*Visit + Age + Years of Education + Presence/Absence of Anti-dementia Drugs as variables.
Time Frame: Baseline, Week 72
Population: All participants in Part B who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
Score on a scale | 1.87 (0.364)

9. Secondary Outcome: Part B: Change From Baseline in Brain Amyloid Plaque Deposition as Measured by Florbetapir F18 Positron Emission Tomography (PET) Scan
Description: Florbetapir PET imaging was used as a quantitative amyloid biomarker. Florbetapir PET scans at baseline and at 36 weeks after the first treatment were used to quantitatively estimate change in amyloid plaques. Quantitative amyloid burden was first formalized as the average Standardized Uptake Value Ratio (SUVR) in six predetermined cortical areas of the brain relative to the cerebellum as a reference region. Larger SUVR reflects the larger cortical amyloid burden relative to cerebellum. SUVR values were further calibrated to a centiloid (CL) scale. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. LS Mean was determined by ANCOVA model using originating study's Baseline + Age + Treatment (Type III sum of squares) as variables.
Time Frame: Baseline, Week 36
Population: All participants in Part B, who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Centiloids
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 36
Centiloids | -80.1 (4.40)

10. Secondary Outcome: Part B: Change From Baseline in Whole Brain Volume as Measured by Volumetric Magnetic Resonance Imaging (vMRI)
Description: Change from Baseline in Whole Brain Volume as Measured by vMRI in Part B. LS mean were derived using MMRM model with fixed factors for visit, and covariates for baseline score, and age at baseline.
Time Frame: Baseline, Week 72
Population: All participants in Part B who received at least one dose of donanemab and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeters (cm3)
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 55
cubic centimeters (cm3) | -27.75 (2.060)

11. Secondary Outcome: Part B: Pharmacokinetics (PK): Trough Concentrations of Donanemab (Ctrough)
Description: PK: Trough Concentration of donanemab. Ctrough is the concentration of drug in the blood immediately before the next dose of drug was administered.
Time Frame: Predose at Week 8 and Week 16
Population: All participants in Part B, who received at least one dose of donanemab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 53
micrograms per milliliter (μg/mL)
  Ctrough at Week 8 | 5.62 (165)
  Ctrough at Week 16: number analyzed (Participants) | 39
  Ctrough at Week 16 | 6.64 (581)

12. Secondary Outcome: Part B: Number or Participants With Treatment-Emergent Anti-Drug Antibodies (TE ADA) of Donanemab
Description: Number of participants in Part B with positive Anti-drug antibodies (TE ADA+) was reported. A TE ADA evaluable participant is classified as TE ADA+ if they have at least one postbaseline titer that is 4 times or more higher than the baseline titer (treatment-boosted). If the baseline result is ADA Not Present, the subject is considered TE ADA+ if there is at least one postbaseline result showing ADA present with a titer of 1:10 or higher (treatment-induced).
Time Frame: Baseline, 4, 8, 16, 24, 36, 48, 60, 72, 84, and 96 Weeks
Population: All participants in Part B who received at least one dose of donanemab and had baseline and at least one post baseline ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Donanemab
Number analyzed (Participants) | 47
Participants | 38

ADVERSE EVENTS:
Time Frame: Baseline Up To 96 Weeks
Description: All enrolled participants. Participants in Part A did not receive any intervention (i.e., study drug). As such, there were no treatment emergent adverse events in Part A. Per pre-planned analysis, adverse events for Part A were reported as per the groups they were randomized into (Group 1 and Group 2) and not as per VTC or on-site as every participant was supposed to participate in both VTC and on-site assessments.
Groups:
- Period 1: Part A - Group 1: Validation of Remote Scale Assessments: Participants from the originating trials did not receive any drug in Part A. Participants in Group 1 underwent cognitive/functional scale assessment at the study site (on-site), followed by an at-home assessment (VTC; video teleconference).
- Period 1: Part A - Group 2: Validation of Remote Scale Assessments: Participants from the originating trials did not receive any drug in Part A. Participants in Group 2 underwent cognitive/functional scale assessment at home (VTC), followed by assessment on-site.
- Period 2: Part B: Donanemab: Participants who had received placebo in the originating trials received 700 mg donanemab administered IV Q4W for 3 doses, then 1400 mg donanemab administered IV Q4W for up to 48 weeks.
Arm/Group | Period 1: Part A - Group 1: Validation of Remote Scale Assessments | Period 1: Part A - Group 2: Validation of Remote Scale Assessments | Period 2: Part B: Donanemab
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/45 | 2/55
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/45 | 16/55
Other Adverse Events (participants affected / at risk) | 0/50 | 0/45 | 40/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Part A - Group 1: Validation of Remote Scale Assessments (N=50) | Period 1: Part A - Group 2: Validation of Remote Scale Assessments (N=45) | Period 2: Part B: Donanemab (N=55)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Part A - Group 1: Validation of Remote Scale Assessments (N=50) | Period 1: Part A - Group 2: Validation of Remote Scale Assessments (N=45) | Period 2: Part B: Donanemab (N=55)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (16)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 7 (10)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 8 (15)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 0 (0) | 0 (0) | 10 (10)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 (0) | 0 (0) | 15 (16)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Superficial siderosis of central nervous system (Nervous system disorders) | 0 (0) | 0 (0) | 3 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT04640077/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT04640077/SAP_001.pdf